CLINICAL TRIAL: NCT00353431
Title: Evaluation of an Algorithm for Intensive s.c. Insulin Therapy in Emergency Room Patients With Hyperglycaemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EKBB13/06; ISRCTN55224894 (Registry Identifier: Current Controlled Trials Database)
Record Dates: First submitted 2006-07-17; First posted 2006-07-18 (Estimated); Results first posted 2012-05-08 (Estimated); Last update posted 2012-05-18 (Estimated); Status verified 2012-05

CONDITIONS: Hyperglycemias
Keywords: Hyperglycaemia; algorithm; emergency; s.c. insulin therapy; Emergency patient
MeSH Terms: conditions — Hyperglycemia; Emergencies | interventions — Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Conventional insulin group:
  In the conventional insulin group only the meal-glucose adapted sliding scale at beginning is pre-determined. All adaptations of the insulin sliding scale remain upon the discretion of the treating physician.
  Interventions: Drug: Novorapid ®, Novo Nordisk, Denmark
- 2 (Experimental): Intensive insulin therapy algorithm:
  The algorithm in the intensive insulin group contains four insulin resistance factors, depending on baseline features of the patients and on the changes of plasma glucose levels after insulin administration. Every two to four hours the plasma glucose level is measured and Insulin aspart (Novorapid®) is injected s.c. according to the scheme. If the patient is eating, the dose of Insulin aspart (NovoRapid®)is increased according to the amount of carbohydrate intake.
  Interventions: Drug: Novorapid ®, Novo Nordisk, Denmark

INTERVENTIONS:
Drug: Novorapid ®, Novo Nordisk, Denmark — Comparison of a sliding scale with an intensive s.c. scale
  Other Names: insulin aspart,; Novolog

SUMMARY:
The aim of this study is to test the safety and efficacy of a new algorithm for intensive s.c. insulin injection in medical emergency patients with hyperglycaemia (plasma glucose concentration ≥ 8 mmol/l)

DETAILED DESCRIPTION:
BACKGROUND: Prospective randomized trials have shown that near-normoglycemic blood glucose control using insulin infusions achieves a significant reduction in mortality of severely ill patients in intensive care units, of patients with acute myocardial infarction and with stroke. This implies that most severely ill patients with hyperglycemia should be treated with insulin to reach near-normoglycemia. However, this is not common practice today in emergency room admissions outside the intensive care unit, and strategies to achieve near-normoglycemia safely outside the ICU setting with s.c. injections (insulin infusions are too risky outside the ICU) have not been established.

AIM: To evaluate an insulin therapy algorithm using s.c. injections which permits effective and safe glycemic management of emergency room patients with hyperglycemia.

DESIGN: Randomized, controlled trial with an open intervention. Patients presenting with hyperglycemia on admission to the emergency room are randomized 1:1 either to conventional treatment (conventional insulin group) or to intensive treatment (intensive insulin group).

METHODS: 140 patients admitted to the medical emergency rooms of the University Hospital Basel and the Regional Hospital of Solothurn will be included and randomized as described above. All patients with plasma glucose levels exceeding 8.0 mmol/l will be included.

Exclusion criteria include severely immunocompromised patients, patients in shock, patients with terminal illnesses on palliative care, type 1 diabetes with or without ketoacidosis and patients which require intensive care unit (ICU) or cardial care unit (CCU) therapy.

PRIMARY ENDPOINT: Time in the glycaemic target range (5.5-7.0 mmol/l) during the period of observation of 48 hours (expected to be longer in the intensive insulin group)

SECONDARY ENDPOINTS: Time to reach the target range. Frequency of hypoglycaemia (plasma glucose < 3.8 mmol/l). Frequency of severe hypoglycaemia (plasma glucose < 2.5 mmol/l. Frequency of hypokalaemia.

ELIGIBILITY:
Inclusion Criteria:

* all patients with hyperglycaemia (≥ 8.0 mmol/l) admitted to the medical emergency room.
* patients with presumed hospitalisation in ER or medical ward of more than 48 h duration.

Exclusion Criteria:

* patients in shock (defined as hypotension or shock index > 1 with oliguria, changed mental status and metabolic acidosis)
* patients with a terminal illness on palliative care
* patients with type 1 diabetes
* patients with insulin pump therapy
* patients with need for hospitalisation in the intensive or coronary care unit.
* patients with presumed hospitalisation shorter than 48 hours
* known pregnancy (in women with childbearing potential pregnancy test for exclusion mandatory)
* no informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2006-12; Primary Completion 2010-04 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Keller, MD, Prof, Principal Investigator — Division of Endocrinology, Diabetes & Clinical Nutrition, Dept of Internal Medicine
Locations (1):
- Division of Endocrinology, Diabetes & Clinical Nutrition, Dept of Internal Medicine,, Basel, Canton of Basel-City, Switzerland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Basel 22.01.2007 until 31.08.2008 Recruitment Solothurn 30.12.2006-29.04.2010
Groups:
- Conventional Insulin Group: In the conventional insulin group only the meal-glucose adapted sliding scale at beginning is pre-determined. All adaptations of the insulin sliding scale remain upon the discretion of the treating physician.
- Intensive Insulin Therapy Algorithm: The algorithm in the intensive insulin group contains four insulin resistance factors, depending on baseline features of the patients and on the changes of plasma glucose levels after insulin administration. Every two to four hours the plasma glucose level is measured and Insulin aspart (Novorapid®) is injected s.c. according to the scheme. If the patient is eating, the dose of Insulin aspart (NovoRapid®)is increased according to the amount of carbohydrate intake.
Period: Overall Study
Arm/Group | Conventional Insulin Group | Intensive Insulin Therapy Algorithm
Started | 63 | 67
Completed | 63 | 67
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional Insulin Group | Intensive Insulin Therapy Algorithm | Total
Number analyzed (Participants) | 63 | 67 | 130
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 15 | 26
  >=65 years | 52 | 52 | 104
Age Continuous [Mean (Standard Deviation); unit: years] | 74.22 (8.77) | 72.43 (11.67) | 73.30 (10.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 29 | 63
  Male | 29 | 38 | 67
Region of Enrollment [Number; unit: participants]
  Switzerland | 63 | 67 | 130

OUTCOME MEASURES:

1. Primary Outcome: Time in the Glycaemic Target Range (5.5-7.0 mmol/l) During the Period of Observation of 48 Hours
Description: Hours in which the plasma glucose was between 5.5 and 7.0 mmol/l (expected to be longer in the intensive insulin group)
Time Frame: 48 h
Population: Intension to treat
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Conventional Insulin Group | Intensive Insulin Therapy Algorithm
Number analyzed (Participants) | 63 | 67
hours | 13.0 (14.7) | 22.5 (10.5)

2. Secondary Outcome: Time to Reach the Target Range
Description: Hours needed to reach 5.5.-7.0 mmol/l (expected to be shorter in the intensive insulin group).
Time Frame: 24 h
Population: Intension to treat
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Conventional Insulin Group | Intensive Insulin Therapy Algorithm
Number analyzed (Participants) | 63 | 67
hours | 24.3 (18.4) | 11.8 (9.4)

3. Secondary Outcome: Frequency of Hypoglycemia
Description: absolute number of participants with hypoglycemia (plasma glucose < 3.8 mmol/l) (safety endpoint, expected to be similar in the two groups)
Time Frame: during observation of 48 hours
Measure: Number; unit: participants
Arm/Group | Conventional Insulin Group | Intensive Insulin Therapy Algorithm
Number analyzed (Participants) | 63 | 67
participants | 4 | 13

4. Secondary Outcome: Frequency of Severe Hypoglycaemia
Description: Number of participants with severe hypoglycaemia (plasma glucose < 2.5 mmol/l) (safety endpoint, expected to be similar in the two groups)
Time Frame: during observation of 48 hours
Measure: Number; unit: participants
Arm/Group | Conventional Insulin Group | Intensive Insulin Therapy Algorithm
Number analyzed (Participants) | 63 | 67
participants | 0 (0) | 1 (0)

5. Secondary Outcome: Frequency of Hypokalaemia
Description: Number of participants with hypokalaemia (potassium < 3.6 mmol/l, safety endpoint, expected to be similar in the two groups)
Time Frame: during observation of 48 hours
Measure: Number; unit: participants
Arm/Group | Conventional Insulin Group | Intensive Insulin Therapy Algorithm
Number analyzed (Participants) | 63 | 67
participants | 15 | 15

ADVERSE EVENTS:
Time Frame: 48 h
Description: Adverse event as Hypoglycaemia and hypokalemia Serious adverse events were death or immediate risk of death
Arm/Group | Conventional Insulin Group | Intensive Insulin Therapy Algorithm
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/67
Other Adverse Events (participants affected / at risk) | 18/63 | 26/67
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional Insulin Group (N=63) | Intensive Insulin Therapy Algorithm (N=67)
Hypokalemia (Metabolism and nutrition disorders) | 15 (15) | 15 (15) — Blood samples at admission, day 1 und day 2
Hypoglycemia (Metabolism and nutrition disorders) | 3 (4) | 11 (14) — Blood glucose measurements according the protocol

LIMITATIONS AND CAVEATS:
Small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes